CLINICAL TRIAL: NCT04094675
Title: Sirolimus for Cowden Syndrome With Colon Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: PTEN Research (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Peter P Stanich, Associate Professor, Division of Gastroenterology, Hepatology & Nutrition, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0179
Record Dates: First submitted 2019-05-13; First posted 2019-09-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: PTEN Gene Mutation; PTEN Hamartoma Tumor Syndrome; PTEN Hamartoma Syndrome; Cowden Syndrome; Bannayan Syndrome; Bannayan Zonana Syndrome; Polyposis
Keywords: PTEN; Cowden syndrome; PHTS; Colon polyposis; sirolimus; Rapamycin; mTOR inhibitor
MeSH Terms: conditions — Hamartoma Syndrome, Multiple | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Open-label pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): There will be a clinic visit and colonoscopy at study entrance with standard of care sampling and assessment of polyps, including resection of concerning polyps. The investigators will also collect data on well-being via the SF-36 health survey (a validated questionnaire to help monitor this aspect given anecdotal patient-level reports of improvement while on therapy).
  Study subjects will then begin sirolimus 2 mg by mouth daily for 1 year.
  Laboratories will be checked at 4 days after initiation, at 2 weeks after initiation, then every 4 weeks for 3 months, then every 3 months to complete the year of therapy
  Participants will have a clinic visit at 3, 6 and 9 months and include well-being assessment with the SF-36 health survey.
  Participants will have a clinic visit with well-being assessment and perform colonoscopy at study closure at 12 months. The investigators will perform standard of care sampling and assessment of polyps, including resection of concerning polyps.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Use of sirolimus 2 mg by mouth daily for 1 year
  Other Names: Rapamycin; Rapamune

SUMMARY:
Colon polyposis (the presence of multiple colon polyps) is very common with Cowden syndrome, as over 60% of patients have 50 or more polyps. In a previous clinical trial, some participants had reduction in the number of colon polyps with the use of the medication sirolimus for a very short time period. This study is investigating sirolimus and its effect on the number of colon polyps in patients with Cowden syndrome and polyposis over a 1 year period.

DETAILED DESCRIPTION:
PTEN is a tumor suppressor gene that regulates the cell cycle through the phosphoinositide 3-kinase (PI3K)/Akt/mTOR pathway. When germline mutations in PTEN occur, the result is Cowden syndrome (or less commonly one of several related disorders collectively called the PTEN hamartoma tumor syndrome). This is characterized by the growth of hamartomas and a high risk of cancer in multiple organ systems. This includes colon polyps in 92.5% of Cowden syndrome patients and 64% with an estimated 50 or more polyps. Although outcomes of this are under reported, series suggest 20-38% of patients will receive colectomy.

Current clinical practice for Cowden syndrome is based on close surveillance for the development of cancers. Sirolimus (also known as rapamycin) is a specific inhibitor of mTOR that is FDA-approved for immunosuppression and use in several types of cancers as chemotherapy. It has also been used successfully in other hamartomatous syndromes including lymphangioleiomyomatosis. There is also a completed pilot clinical trial for adults with Cowden syndrome in which some had reduction in the number of colon polyps with the use of the medication sirolimus for a very short time period.

This will be an open-label pilot trial to determine whether sirolimus reduces colon polyp burden in Cowden syndrome. Sirolimus will be administered for one year. Colonoscopy with polyp estimation will be performed at trial entrance and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Cowden syndrome or other PTEN hamartoma tumor syndrome spectrum disorder
* Confirmed pathogenic or likely pathogenic PTEN germline mutation on genetic testing
* Previous colonoscopy with colon polyposis. This is defined for the study as either too many polyps to remove endoscopically as judged by the performing physician at the last colonoscopy or findings indicating at least an InSIGHT stage 1 score (over 20 polyps).
* Age 18 or greater
* Capacity to consent to study

Exclusion Criteria:

* Pregnancy or plans for pregnancy while on treatment or within 3 months of stopping treatment (for both women and men)
* Chronic kidney disease
* Chronic renal disease
* History of colon cancer or colon adenoma with high grade dysplasia
* History of colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in colon polyp burden by number | 1 year
  Assessment of change in number of colon polyps. This will be assessed for each segment of colon (ascending, transverse, descending, sigmoid, rectum) and then aggregated into a total number of colon polyps. The entrance result will be compared to the final result for each participant.
Change in colon polyp burden by staging | 1 year
  Assessment of change in staging of colon polyps by using the International Society for Gastrointestinal Hereditary Tumors (InSIGHT) polyposis staging system. The InSight staging system divides colorectal polyposis into 5 progressive stages based on polyp number and size (Stage 0: <20 polyps, all <5 mm; Stage 1: 20-200 polyps, most <5 mm, none, >1 cm; Stage 2: 200-500 polyps, <10 that are >1 cm; Stage 3: 500-1000 polyps or any number if there are 10-50 that are >1 cm and amenable to complete polypectomy; Stage 4: >1000 polyps and/or any polyps grown to confluence and not amenable to simple polypectomy; any high-grade dysplasia or invasive cancer). The entrance result will be compared to the final result for each participant.

SECONDARY OUTCOMES:
Change in well-being assessment | 1 year
  Assessment in change in overall health and quality of life as quantified by the SF-36 (Short Form) Health Survey. The SF-36 is a widely-used and standardized survey of participant responses to 36 questions that measures health-related quality of life. Each question has answers that are given a correlating score from 0 to 100, with a high score representing a more favorable health state. Through the combination of specific questions and averaging the scores, there are 8 scales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality, mental health, social functioning, bodily pain, and general health) that are reported with scores from 0 to 100, with a high score representing a more favorable health state. These can also be averaged into a physical component summary score and mental component summary score that is again from 0 to 100, with a high score representing a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Stanich, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanich PP, Pilarski R, Rock J, Frankel WL, El-Dika S, Meyer MM. Colonic manifestations of PTEN hamartoma tumor syndrome: case series and systematic review. World J Gastroenterol. 2014 Feb 21;20(7):1833-8. doi: 10.3748/wjg.v20.i7.1833. PMID 24587660
- [Background] Stanich PP, Owens VL, Sweetser S, Khambatta S, Smyrk TC, Richardson RL, Goetz MP, Patnaik MM. Colonic polyposis and neoplasia in Cowden syndrome. Mayo Clin Proc. 2011 Jun;86(6):489-92. doi: 10.4065/mcp.2010.0816. PMID 21628613
- [Background] Heald B, Mester J, Rybicki L, Orloff MS, Burke CA, Eng C. Frequent gastrointestinal polyps and colorectal adenocarcinomas in a prospective series of PTEN mutation carriers. Gastroenterology. 2010 Dec;139(6):1927-33. doi: 10.1053/j.gastro.2010.06.061. Epub 2010 Jun 27. PMID 20600018
- [Background] Komiya T, Blumenthal GM, DeChowdhury R, Fioravanti S, Ballas MS, Morris J, Hornyak TJ, Wank S, Hewitt SM, Morrow B, Memmott RM, Rajan A, Dennis PA. A Pilot Study of Sirolimus in Subjects with Cowden Syndrome or Other Syndromes Characterized by Germline Mutations in PTEN. Oncologist. 2019 Dec;24(12):1510-e1265. doi: 10.1634/theoncologist.2019-0514. Epub 2019 Jul 26. PMID 31350329
- [Background] Lynch PM, Morris JS, Wen S, Advani SM, Ross W, Chang GJ, Rodriguez-Bigas M, Raju GS, Ricciardiello L, Iwama T, Rossi BM, Pellise M, Stoffel E, Wise PE, Bertario L, Saunders B, Burt R, Belluzzi A, Ahnen D, Matsubara N, Bulow S, Jespersen N, Clark SK, Erdman SH, Markowitz AJ, Bernstein I, De Haas N, Syngal S, Moeslein G. A proposed staging system and stage-specific interventions for familial adenomatous polyposis. Gastrointest Endosc. 2016 Jul;84(1):115-125.e4. doi: 10.1016/j.gie.2015.12.029. Epub 2016 Jan 6. PMID 26769407
- [Derived] Stanich PP, Gofar K, Roberts ME, Hussan H. Sirolimus for Colon Polyposis in PTEN Hamartoma Tumor Syndrome. Clin Transl Gastroenterol. 2025 Jun 6;16(8):e00871. doi: 10.14309/ctg.0000000000000871. eCollection 2025 Aug 1. PMID 40478255

DOCUMENTS (1):
  • Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT04094675/ICF_001.pdf